CLINICAL TRIAL: NCT06997367
Title: A Phase II, Randomized, Double-blind Trial to Assess the Safety and Immunogenicity of MTBVAC (BBV169), With BCG Vaccine as a Comparator in Healthy Adolescent and Adult Populations
Brief Title: Safety and Immunogenicity of a Mycobacterium Tuberculosis Vaccine MTBVAC in Healthy Indian Adults and Adolescents (BBV169/2024)
Acronym: MTBVACph2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BBIL/MTBVAC-II/2024
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis (TB)
Keywords: MTBVAC; BCG; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized trial assessing the safety and immunogenicity of the MTBVAC vaccine, with BCG as a comparator. A total of 164 participants aged 12 to 65 will be randomized in a 1:1 ratio to receive a single intradermal dose of either MTBVAC or BCG on Study Day 0. Participants will be split into two cohorts based on QFT-Plus assay results (negative and positive), with each cohort including 82 QFT participants.
  Group I (Age: ≥ 18 years): 10 adults per cohort will be enrolled and safety reviewed by the Data and Safety Monitoring Board (DSMB) two weeks post-vaccination before recruiting more adults and participants aged 12 to <18.
  Group II (Age: ≥ 12 to <18 years): After initial adult recruitment, 10 participants per cohort aged 12 to <18 will be enrolled, also reviewed by the DSMB. The study aims to ensure that at least 20% of participants in both arms are adolescents.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The trial participant, trial investigator, and sponsor will be blinded to the intervention given. The pharmacist will be unblinded staff in the trial and will not be the part of any other trial procedures or collection of safety information.
  Test and control vaccines will be packed into identical white cartons with only kit numbers. On the day of dosing, the unblinded pharmacist at each trial site will be provided with the required participant information.The pharmacist will prepare and dispense the injection as per the randomization code(under physical partition for maintaining blinding) and provide the syringe to the trialnurse to administer the IP to the participant.The Data and Safety Monitoring Board (DSMB) will receive aggregate data for safetyreview. If necessary, data may be unblinded to individual participant treatment assignments to adequately assess safety issues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTBVAC (Experimental): Biological: MTBVAC (BBV169) Mycobacterium tuberculosis vaccine
  Interventions: Biological: MTBVAC
- BCG (Active Comparator): Biological: BCG [TUBERVAC]
  Interventions: Biological: BCG Sii

INTERVENTIONS:
Biological: MTBVAC — MTBVAC (BBV169) vaccine is a freeze-dried powder containing live attenuated Mycobacterium tuberculosis (M. tb), which is presented as a lyophilized product in a 10- dose vial. After reconstitution with 1.0 mL sterile water for injection, one dose (0.1mL) of vaccine contains 5 x10^5 CFU live attenuated M. tb. One dose (0.1mL) of the MTBVAC (BBV169) vaccine is to be administered in the right deltoid region via the intradermal route.
  Other Names: BBV169
  Arms: MTBVAC
Biological: BCG Sii — Comparator vaccine: BCG Vaccine (TUBERVAC- Moscow strain), manufactured by Serum Institute of India, is a freeze-dried powder containing an attenuated strain of Bacillus Calmette-Guerin Mycobacterium bovis as a lyophilized product in a 10-dose vial. After reconstitution with 1.0 mL diluent (Sodium chloride) for injection, one dose (0.1mL) of BCG vaccine will be administered in the right deltoid region via the intradermal route.
  Arms: BCG

SUMMARY:
Phase II trial to establish the safety, reactogenicity, and immunogenicity of the MTBVAC with a licensed BCG vaccine as a comparator in both TB naïve (QFT PLUS negative) and TB exposed (QFT PLUS positive) healthy adults and adolescents.

DETAILED DESCRIPTION:
Phase II, double-blind, randomized, safety and immunogenicity trial with BCG vaccine as a comparator in 164 healthy adults and adolescents and with both positive and negative interferon gamma release assay (IGRA) test result.

Objective: To evaluate the immunogenicity of MTBVAC compared to BCG in all participants using PBMC Participants meeting the inclusion and exclusion criteria will be randomized within a study cohort in a 1:1 ratio to receive a single dose of MTBVAC or BCG vaccine administered intradermally. Only HIV-negative participants will be eligible for enrolment. A total of 164 participants aged 12-65 years will be enrolled into one of two cohorts based on their based on the QFT-Plus assay results (QFT negative and QFT positive).

Cohort 1 will include 82 QFT Negative participants Cohort 2 will include 82 QFT Positive participants. Study participants will be randomized in a 1:1 ratio within each cohort to receive MTBVAC (Total N=82, includes 41 QFT negative & 41 QFT positive participants) or BCG (Total N=82, includes 41 QFT negative & 41 QFT positive participants) Participants will be followed up for safety and Immunogenicity following vaccination via regular visits.

At least 20% of the participants will be the adolescent population in each cohort in treatment and comparator arms.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and informed Assent from Adolescents
2. Participants of either gender of age between ≥12 to ≤65 years at the time of obtaining informed consent/assent.
3. Good general health as determined by the discretion of the investigator (vital signs, medical history, and physical examination).
4. Expressed interest and Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
5. For a female participant of childbearing potential, planning to avoid pregnancy (use of an effective method of contraception or abstinence) from the time of study enrolment until at least three months after IP administration.
6. Male participants of reproductive potential: Willing to use condoms to ensure effective contraception with the female partner from IP administration until three months.
7. No evidence of active TB disease during screening - As confirmed by normal chest radiograph and no sputum positivity by NAAT test for M. tb
8. A negative urine pregnancy test for female participants of childbearing potential.
9. Only participants who are HIV negative 10. Non-diabetic participants with RBS less than 140 mg/dl and as confirmed by medical history

11. Had BCG vaccination, documented through the presence of scar.

Exclusion Criteria:

1. Any chronic febrile illness with oral temperature > 100.4°F on the day of randomization.
2. Clinical evidence of pulmonary pathology.
3. History of any form of TB Disease.
4. Prior or present anti-TB treatment
5. Received Tuberculin Skin Test (TST) within three months (90 days) prior to Study Day 0.
6. Clinical Evidence of Active TB
7. Participants with household contacts of patients with active TB disease
8. History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations (any vaccine).
9. History of allergic disease or reactions.
10. History of previous administration of experimental TB vaccines.
11. Use of any investigational or non-registered product (drug or vaccine) in another experimental protocol other than the trial vaccines within 30 days preceding the vaccination, or planned use during the trial period.
12. Any chronic drug therapy is to be continued during the trial period.
13. Chronic administration of immunosuppressors or other immune-modifying drugs.
14. Administration of any immunoglobulins, any immunotherapy, and/or any blood products within the three months preceding the vaccination or planned administrations during the trial period.
15. Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
16. Participants who are HIV Positive or on ART.
17. Participants with a medical history of diabetes or those whose RBS levels exceed 140 mg/dL
18. Any condition or history of any acute or chronic illness or medication, which, in the opinion of the Investigator, may interfere with the evaluation of the trial objectives.
19. A family history of congenital or hereditary immunodeficiency
20. History of any neurologic disorders or seizures.
21. History of chronic alcohol consumption and/or drug abuse.
22. Congenital defects in the cardiopulmonary and neurological system
23. Pregnant or lactating female.
24. Females who are planning to become pregnant or planning to discontinue contraceptive precautions during the trial period.
25. Those who have been vaccinated with live attenuated vaccines within 30 days of trial vaccine administration and those who are planning to take live attenuated vaccine within 30 days after trial vaccine administration.
26. Administration of any vaccines that are not live attenuated within 30 days before trial vaccine administration.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of MTBVAC compared to BCG in all participants using PBMC | Day 1 through Day 180
  Antigen-specific CD4 response - Frequencies and co-expression patterns of CD4 cells expressing IFN-γ, and/or TNF, and/or IL-2, induced by MTBVAC and BCG measured on Day 0, 28, 56, 90 and 180 using PBMC Intracellular cytokine assay

SECONDARY OUTCOMES:
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- Immediate adverse events | 30 minutes of vaccination
  Occurrence of immediate adverse events within 30 minutes of vaccination
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- Solicited adverse events | Day 1 through Day 14
  Occurrence of Solicited adverse events within fourteen days of vaccination
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- Injection site reactions | Day 1 through Day 90
  Injection site reactions will be followed-up for 90 days.
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- Unsolicited adverse events | Day 1 through Day 360
  Occurrence of any unsolicited adverse events throughout the study duration
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- Serious adverse events (SAE s) | Day 1 through Day 360
  Occurrence of serious adverse events (SAEs)
To evaluate the safety and reactogenicity of MTBVAC compared to BCG- AESI (Adverse Event of Special Interest) | Day 1 through Day 360
  AESI (Adverse Event of Special Interest) is to be considered throughout the trial period.

OTHER OUTCOMES:
To evaluate QFT conversion and reversion rates in QFT-negative adults and adolescents | Day 1 through Day 180
  Qualitative (positive or negative)
Humoral immune response in all participants | Day 1 through Day 180
  Serum IgG Antibodies- Evaluate humoral immune response at Days 0, 28, 56, 90 and 180
To assess the immunogenicity of MTBVAC compared to BCG using WBA at one site | Day 1 through Day 180
  Antigen-specific secretory cytokine responses - Evaluate secretory cytokine responses post stimulation by TB specific antigens, measured on - Day 0, 28, 56, 90, and 180 using whole blood intracellular cytokine assay at one site.
To assess Antigen-specific CD8 response of MTBVAC compared to BCG | Day 1 through Day 180
  Antigen-specific CD8 response: Frequencies and co-expression patterns of CD8 cells expressing IFN-γ, and/or TNF, and/or IL-2, induced by MTBVAC and BCG measured on Day 0, 28, 56, 90 and 180 using PBMC Intracellular cytokine assay at all sites
To evaluate QFT conversion and reversion rates in QFT-negative adults and adolescents | Day 1 through Day 180
  Quantitative (TB Ag-Nil, IFN-γ concentration) QuantiFERON -Gold Plus assay results.
  QuantiFERON conversion will be defined as a positive test without a prior positive test; QuantiFERON reversion will be defined as a negative test following a positive test). QFT will be done on Day 28, 56, 90, and 180.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.V.Krishna Mohan, PhD, Study Director — Bharat Biotech International Limited
Locations (2):
- India (2):
  - Guru Teg Bahadur Hospital, Delhi
  - AIIMS-Delhi, New Delhi